CLINICAL TRIAL: NCT02724956
Title: Randomized Comparison of Ambu AuraGain and Teleflex Protector Using Clinical and Fiberoptic Assessments in Elective Patients
Brief Title: Ambu AuraGain and Teleflex LMA Protector Fiberoptic Assessments in Elective Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Ambu A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2017-0449; HSC-MS-14-0970 (Other: Previous University of Texas Health Science Center ID)
Record Dates: First submitted 2016-03-22; First posted 2016-03-31 (Estimated); Results first posted 2021-08-31 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-08

CONDITIONS: Anesthesia
Keywords: supraglottic airway device (SGAD) insertion; SGAD; ventilation and intubation; gastric drainage channel; fiberoptic assessment
MeSH Terms: conditions — Respiratory Aspiration | interventions — Laryngeal Masks

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Ambu AuraGain (Experimental): SGAD placement using Ambu AuraGain
  * Lubricate airway tube of SGAD & pass the aScope through until visualization of the carina.
  * Standard Parker Flex Tip endotracheal tube (ETT) size 6.0, 7.0, and 8.0 mm ETT will be used as per anesthesiologist preference.
  * Pass ETT tube down the insertion cord of the Ambu aScope & verify placement.
  * Inflate cuff and remove aScope.
  Interventions: Device: Ambu AuraGain; Device: Ambu aScope
- Teleflex LMA Protector (Experimental): SGAD placement using the Teleflex LMA Protector
  * Lubricate airway tube of SGAD & pass the aScope through until visualization of the carina.
  * Standard Parker Flex Tip ETT size 6.0 and 7.0 mm. ETT will be used as per anesthesiologist preference.
  * Pass ETT tube down the insertion cord of the Ambu aScope & verify placement.
  * Inflate cuff and remove aScope.
  Interventions: Device: Teleflex LMA Protector; Device: Ambu aScope

INTERVENTIONS:
Device: Ambu AuraGain — Pre-curved, rigid airway tube, SGAD. Third generation Ambu laryngeal mask satisfying 3 fundamental airway management needs by integrating gastric access and intubation capability in an anatomically curved single-use device that facilitates rapid establishment of a safe airway. A SGAD used for ventilation, and a conduit for intubation. SGAD insertion followed by fiber-optic evaluation using Ambu aScope.
  Other Names: Supraglottic airway device; SGAD
  Arms: Ambu AuraGain
Device: Teleflex LMA Protector — Pre-curved, rigid airway tube, SGAD: A next-generation, single-use laryngeal mask with a dual gastric drainage channel and pharyngeal chamber. A SGAD used for ventilation, and a conduit for intubation. SGAD insertion followed by fiber-optic evaluation using Ambu aScope.
  Other Names: LMA® Protector™; Supraglottic airway device; SGAD; LMA; laryngeal mask airway
  Arms: Teleflex LMA Protector
Device: Ambu aScope — Flexible scope which will be introduced into airway tube and guided through the SGAD until it will be possible to view the vocal cords. Description of the maximal optical view will be measured by the Percentage of Glottic Opening (POGO).
  Other Names: Ambu® aScope™ 3 Slim

SUMMARY:
Participant is being asked to take part in this study because participant is going to have surgery that requires general anesthesia (in which participant is unconscious for the procedure).

During surgery, anesthesiologists often place a supraglottic airway device (SGAD). An SGAD is a device that helps participant breathe and may help the anesthesiologist put a breathing tube in participant's airway while participant is asleep during surgery. There are many different kinds of SGADs that are readily available for use by anesthesiologists during surgery. The SGADs that are being studied are the Ambu Auragain and the Teleflex LMA Protector.

The goal of this clinical research study is to compare the effectiveness of both devices.

This is an investigational study. Both of the SGADs that are being used on this study are FDA approved and are frequently used for the surgery that participant is going to have. It is investigational to compare the 2 devices.

Up to 50 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Surgery:

Participant will sign a separate consent form for surgery that describes the procedure and its risks. Participant will receive anesthesia through a catheter (sterile flexible tube) in one of participant's veins. During the procedure, participant's vital signs (heart rate, blood pressure, oxygen levels) will be monitored.

Study Groups:

If participant agrees to take part in this study, demographic information (such as participant's age, sex, and race) will be collected.

Participant will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. This is done because no one knows if one study group is better, the same, or worse than the other group. Participant will have an equal (50/50) chance of being assigned to either group. One group will use the Ambu Auragain, and the other will use the Teleflex LMA Protector.

Study Procedures:

After general anesthesia is given and participant falls asleep, the anesthesiologist will place the SGAD. The study staff will measure how easy it is to place the SGAD and how long each different step of the placement takes. Correct placement of the SGAD will be checked using a device with a small camera to help the doctor see participant's airway on a screen. A gastric tube will be placed to measure the volume of air and content of the stomach. Additionally the study doctor may place a breathing tube using the SGAD to make sure air is moving in and out of participant's lungs.

Participant will then be positioned and prepared for the surgery. The study staff will be collecting information from the time participant enters the operating room until the time participant leaves.

Additionally, participant will be interviewed after participant's surgery in the recovery room once participant is awake. Participant will be asked about any pain or soreness participant has, as well as any difficulty breathing, swallowing, or talking. This interview may take up to 5 minutes. Participation in the study will be over after the interview.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years of age or older
2. Scheduled for an elective surgery requiring general anesthesia
3. Scheduled surgery < 4hrs
4. American Society of Anesthesiology (ASA) Physical Status I-III
5. Body Mass Index (BMI) < 30 kg/m2
6. Mallampati I-III
7. Able to bite upper lip via Upper Lip Bite Test (ULBT)
8. Inter-incisor distance > 2.5cm
9. Thyromental distance > 6cm
10. Full range of motion in the neck
11. Has provided written informed consent

Exclusion Criteria:

1. Under the age of 18 years old
2. ASA IV-V
3. Require prone positioning for surgery
4. Scheduled surgery > 4hrs
5. Liquid only diet < 2hrs and/or solids < 8hrs
6. High risk of regurgitation
7. Exhibits signs of respiratory tract pathology (including a sore throat preoperatively)
8. Mallampati IV
9. Unable to bite upper lip via Upper Lip Bite Test (ULBT)
10. Inter-incisor distance < 2.5cm
11. Thyromental distance < 6cm
12. Limited neck movement
13. Airway pathology/facial abnormality
14. Has been diagnosed with/exhibits any mental neurological disorder/disease/condition that would prevent participation in the study in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carin A Hagberg, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The University of Texas (UT) MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ambu AuraGain | Teleflex LMA Protector
Started | 27 | 26
Completed | 26 | 24
Not Completed | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ambu AuraGain: SGAD placement using Ambu AuraGain
  * Lubricate airway tube of SGAD & pass the aScope through until visualization of the carina.
  * Standard Parker Flex Tip endotracheal tube (ETT) size 6.0, 7.0, and 8.0 mm ETT will be used as per anesthesiologist preference.
  * Pass ETT tube down the insertion cord of the Ambu aScope & verify placement.
  * Inflate cuff and remove aScope.
  Ambu AuraGain: Pre-curved, rigid airway tube, SGAD. Third generation Ambu laryngeal mask satisfying 3 fundamental airway management needs by integrating gastric access and intubation capability in an anatomically curved single-use device that facilitates rapid establishment of a safe airway. A SGAD used for ventilation, and a conduit for intubation. SGAD insertion followed by fiber-optic evaluation using Ambu aScope.
  Ambu aScope: Flexible scope which will be introduced into airway tube and guided through the SGAD until it will be possible to view the vocal cords. Description of the maximal optical view will be measured by the Percentage of Glottic Opening (POGO).
- Teleflex LMA Protector: SGAD placement using the Teleflex LMA Protector
  * Lubricate airway tube of SGAD & pass the aScope through until visualization of the carina.
  * Standard Parker Flex Tip ETT size 6.0 and 7.0 mm. ETT will be used as per anesthesiologist preference.
  * Pass ETT tube down the insertion cord of the Ambu aScope & verify placement.
  * Inflate cuff and remove aScope.
  Teleflex LMA Protector: Pre-curved, rigid airway tube, SGAD: A next-generation, single-use laryngeal mask with a dual gastric drainage channel and pharyngeal chamber. A SGAD used for ventilation, and a conduit for intubation. SGAD insertion followed by fiber-optic evaluation using Ambu aScope.
  Ambu aScope: Flexible scope which will be introduced into airway tube and guided through the SGAD until it will be possible to view the vocal cords. Description of the maximal optical view will be measured by the Percentage of Glottic Opening (POGO).
- Total: Total of all reporting groups
Arm/Group | Ambu AuraGain | Teleflex LMA Protector | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 15 | 35
  >=65 years | 6 | 9 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 39
  Male | 5 | 6 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 26 | 24 | 50
Supraglottic Airway (SGA) Sizes [Count of Participants; unit: Participants] — Size 3: 30-50 kg, Size 4: 50-70 kg, and Size 5: 70-100 kg
  Participants
    SGA Size 3 | 6 | 5 | 11
    SGA Size 4 | 19 | 17 | 36
    SGA Size 5 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: 1st Attempt Success With Supraglottic Airway Devices (SGAD)
Description: Success defined as correct placement of SGAD. 1st Attempt success of SGAD either Ambu AuraGain or Teleflex LMA Protector during insertion and placement into an airway.
Time Frame: from Anesthesia Start to Anesthesia Stop, approximately 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Ambu AuraGain | Teleflex LMA Protector
Number analyzed (Participants) | 26 | 24
Participants
  Successful | 25 | 21
  Unsuccessful | 1 | 3

2. Secondary Outcome: Oropharyngeal Leak Pressure (OLP)
Description: OLP measured by a portable, handheld manometer.
Time Frame: from Anesthesia Start to Anesthesia Stop, approximately 1 hour
Population: 8 participants were not recorded due to protocol deviation
Measure: Median (95% Confidence Interval); unit: cmH2O
Arm/Group | Ambu AuraGain | Teleflex LMA Protector
Number analyzed (Participants) | 21 | 21
cmH2O | 35 [22.00 to 68.00] | 37 [15.00 to 56.20]

3. Secondary Outcome: Number of Participants With a Rate of Successful Intubation and Ventilation
Description: Rate of successful intubation and ventilation by utilizing the SGAD as an intubation conduit guided by the Ambu® aScope™ 3 Slim.
Time Frame: from Anesthesia Start to Anesthesia Stop, approximately 1 hour
Population: 1 participant was not analyzed in the Teleflex LMA Protector Arm due to device failure
Measure: Count of Participants; unit: Participants
Arm/Group | Ambu AuraGain | Teleflex LMA Protector
Number analyzed (Participants) | 26 | 23
Participants
  Successful | 21 | 19
  Unsuccessful | 5 | 4

4. Secondary Outcome: Number of Participants With Ease of SGAD Insertion
Description: Qualitative Assessment scale range of 1-4. (1) Easy; (2) Resistance, (3) Difficult; and (4) Unsuccessful.
Time Frame: from Anesthesia Start to Anesthesia Stop, approximately 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Ambu AuraGain | Teleflex LMA Protector
Number analyzed (Participants) | 26 | 24
Participants
  Easy | 25 | 21
  Resistance | 1 | 2
  Difficult | 0 | 0
  Unsuccessful | 0 | 1

5. Secondary Outcome: Glottic Opening (POGO)
Description: POGO Score of 100% on First Attempt at Device Placement. All participant assessments and observations (clinical data) completed and recorded during the 1st visit
Time Frame: from Anesthesia Start to Anesthesia Stop, approximately 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Ambu AuraGain | Teleflex LMA Protector
Number analyzed (Participants) | 26 | 24
Participants
  POGO- Observed | 26 | 20
  POGO- Not Observed | 0 | 4

6. Secondary Outcome: Functionality of Gastric Tube Placement
Description: Functionality of gastric drainage channel which will be inserted through the appropriate channel of the SGAD.
Time Frame: from Anesthesia Start to Anesthesia Stop, approximately 1 hour
Population: 1 participant was not analyzed in the Teleflex LMA Protector Arm due to device failure
Measure: Count of Participants; unit: Participants
Arm/Group | Ambu AuraGain | Teleflex LMA Protector
Number analyzed (Participants) | 26 | 23
Participants
  Easy | 26 | 16
  Resistance | 0 | 1
  Difficult | 0 | 0
  Unsuccessful | 0 | 6

ADVERSE EVENTS:
Time Frame: during the 1st visit, up to 60 minutes
Description: no reportable AE's/SAE's for this study
Arm/Group | Ambu AuraGain | Teleflex LMA Protector
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT02724956/Prot_SAP_000.pdf